CLINICAL TRIAL: NCT02532049
Title: A Phase Ia Clinical Trial to Assess the Safety, Immunogenicity and Ex-vivo Efficacy of New Plasmodium Falciparum Malaria Vaccine Candidates ChAd63 Pfs-IMX313 Alone and With MVA Pfs25-IMX313
Brief Title: A Clinical Trial to Assess the Safety and Immunogenicity of New Malaria Vaccine Candidates ChAd63 Pfs25-IMX313 and MVA Pfs25-IMX313
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VAC062
Record Dates: First submitted 2015-08-07; First posted 2015-08-25 (Estimated); Last update posted 2017-07-17 (Actual); Status verified 2017-07

CONDITIONS: Malaria
Keywords: Malaria; Vaccine; Immune Response
MeSH Terms: conditions — Malaria | interventions — ChAd63 Pfs25-IMX313 malaria vaccine; MVA Pfs25-IMX313 malaria vaccine

ARMS (4):
- Group 1 (Active Comparator): ChAd63 Pfs25-IMX313 (5x10^9 vp)
  Interventions: Biological: ChAd63 Pfs25-IMX313
- Group 2A (Active Comparator): ChAd63 Pfs25-IMX313 (5x10^10 vp)
  Interventions: Biological: ChAd63 Pfs25-IMX313
- Group 2B (Active Comparator): ChAd63 Pfs25-IMX313 (5x10^10) and MVA Pfs25-IMX313 (1x10^8 pfu) 8 weeks later
  Interventions: Biological: ChAd63 Pfs25-IMX313; Biological: MVA Pfs25-IMX313
- Group 2C (Active Comparator): ChAd63 Pfs25-IMX313 (5x10^10) and MVA Pfs25-IMX313 (2x10^8 pfu) 8 weeks later
  Interventions: Biological: ChAd63 Pfs25-IMX313; Biological: MVA Pfs25-IMX313

INTERVENTIONS:
Biological: ChAd63 Pfs25-IMX313
Biological: MVA Pfs25-IMX313
  Arms: Group 2B; Group 2C

SUMMARY:
This is a clinical trial in which healthy volunteers will be administered one or two experimental malaria vaccines. ChAd Pfs-IMX313 will either be administered alone or with MVA Pfs25-IMX313 in a prime-boost regime.

All vaccines will be administered intramuscularly.

Group 1 will receive one dose of ChAd63 Pfs25-IMX313 at 5x10^9 vp.

Group 2A will receive one dose of ChAd63 Pfs-IMX313 at 5x10^10 vp.

Group 2B will receive one dose of ChAd63 Pfs-IMX313 at 5x10^10 vp and one dose of MVA Pfs25-IMX313 at 1x10^8 pfu eight weeks later.

Group 2C will receive one dose of ChAd63 Pfs25-IMX313 at 5x10^10 vp and one dose of MVA Pfs25-IMX313 at 2x10^8 pfu eight weeks later.

The study will assess the safety of the vaccinations, and the immune responses to the vaccination. Immune responses are measured by tests on blood samples.

Healthy volunteers will be recruited in Oxford and Southampton, England.

ELIGIBILITY:
Inclusion Criteria:

The volunteer must satisfy all the following criteria to be eligible for the study:

* Healthy adults aged 18 to 50 years
* Able and willing (in the Investigator's opinion) to comply with all study requirements
* Willing to allow the investigators to discuss the volunteer's medical history with their General Practitioner
* For females only, willingness to practice continuous effective contraception (see below) during the study and a negative pregnancy test on the day(s) of screening and vaccination
* Agreement to refrain from blood donation during the course of the study
* Provide written informed consent

Exclusion Criteria:

The volunteer may not enter the study if any of the following apply:

* Participation in another research study involving receipt of an investigational product in the 30 days preceding enrolment, or planned use during the study period
* Prior receipt of an investigational malaria vaccine or any other investigational vaccine likely to impact on interpretation of the trial data.
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccine candidate
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled and topical steroids are allowed)
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine, e.g. egg products.
* Any history of anaphylaxis in relation to vaccination
* Pregnancy, lactation or willingness/intention to become pregnant during the study
* History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ)
* History of serious psychiatric condition likely to affect participation in the study
* Any other serious chronic illness requiring hospital specialist supervision
* Suspected or known current alcohol abuse as defined by an alcohol intake of greater than 42 units every week
* Suspected or known injecting drug abuse in the 5 years preceding enrolment
* Seropositive for hepatitis B surface antigen (HBsAg)
* Seropositive for hepatitis C virus (antibodies to HCV)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2015-10-12 (Actual); Primary Completion 2017-05-25 (Actual); Study Completion 2017-05-25 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events | 8 months
  The specific endpoints for safety and reactogenicity will be actively and passively collected data on adverse events.

SECONDARY OUTCOMES:
Immunogenicity of ChAd63 Pfs25-IMX313 when administered to healthy volunteers alone, and with MVA Pfs25-IMX313 in a prime-boost regime. | 8 months
Ex-vivo efficacy of ChAd63 Pfs25-IMX313 when administered to healthy volunteers alone, and with MVA Pfs25-IMX313 in a prime-boost regime. The functional activity of the vaccine induced antibodies will be tested using membrane-feeding assays. | 8 months

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - CCVTM, University of Oxford, Churchill Hospital, Oxford
  - NIHR Wellcome Trust Clinical Research Facility, Southampton

REFERENCES:
- [Derived] de Graaf H, Payne RO, Taylor I, Miura K, Long CA, Elias SC, Zaric M, Minassian AM, Silk SE, Li L, Poulton ID, Baker M, Draper SJ, Gbesemete D, Brendish NJ, Martins F, Marini A, Mekhaiel D, Edwards NJ, Roberts R, Vekemans J, Moyle S, Faust SN, Berrie E, Lawrie AM, Hill F, Hill AVS, Biswas S. Safety and Immunogenicity of ChAd63/MVA Pfs25-IMX313 in a Phase I First-in-Human Trial. Front Immunol. 2021 Jul 14;12:694759. doi: 10.3389/fimmu.2021.694759. eCollection 2021. PMID 34335606